CLINICAL TRIAL: NCT00179556
Title: Daidzein-rich Isoflavone-aglycones for Menopausal Symptoms
Brief Title: Effects of Soy Isoflavones on Menopausal Hot Flashes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Nichimo - Tokyo, Japan (Unknown)
Responsible Party: Principal Investigator, Hope Ricciotti, Associate Professor of Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002P000037
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Menopausal Symptoms
Keywords: Hot flashes; Menopausal symptoms; Soybean germ; Aglycones; Menopause
MeSH Terms: conditions — Hot Flashes

INTERVENTIONS:
Drug: Isoflavone supplement

SUMMARY:
Hot flashes occur in three quarters of menopausal women, and can negatively impact quality of life. Interest has arisen in isoflavones, found in rich supply in soy products, as therapy for hot flashes. The study examines the effect of a new soy supplement, as compared to a placebo, in menopausal women on hot flash symptoms.

DETAILED DESCRIPTION:
Hot flashes occur in 75% of menopausal women and impact quality of life. Interest has arisen in isoflavones, found in rich supply in soy products, as therapy for hot flashes. The effect of a daidzein-rich isoflavone-aglycone supplement from soy germ fermentation with Koji fungus, on the severity and frequency of hot flashes in postmenopausal women is being examined in a randomized, placebo controlled, double-blinded clinical trial. The study is a 13 week trial in which subjects record their hot flash frequency and severity in a diary. Subjects are given 40 mg or 60 mg of isoflavones (or placebo) once a day. This isoflavone-aglycone extract (Agly-Max TM, Nichimo, Shinagawa, Tokyo, Japan) is a product prepared from soybean germ fermentation with Koji fungus (Aspergliius awamori) producing ß-glycosidase efficiency, followed by ethanol and water extraction and purification by using a proprietary extraction procedure. The product is rich in daidzein (70% daidzein, 10% genistein, and 20% glycitein).

ELIGIBILITY:
Inclusion Criteria:

No menstrual period for at least six months, Hot flashes at least four t imes per day, Ages 38-65

Exclusion Criteria:

Pregnant, BMI>45, History of breast cancer or other estrogen dependent tumors, Abnormal uterine bleeding, Heart, renal, or liver disease, Diabetes, Women taking hormone replacement therapy or serotonin reuptake inhibitors, Women taking any dietary supplements for the treatment of hot flashes (ex. soy supplements, vitamin E, flaxseed, red clover extract) within the past 30 days

Ages: 38 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2003-06; Primary Completion 2005-07 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Hot flash frequency and severity

SECONDARY OUTCOMES:
Menopausal quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hope Ricciotti, MD, Principal Investigator — Beth Israel Deaconess Medical Center; George Blackburn, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center; Lalita Khaodhiar, MD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States